CLINICAL TRIAL: NCT00727103
Title: Varenicline Treatment in Alcohol and Nicotine Dependent Patients With Schizophrenia - a Double Blind, Placebo Controlled Trial
Brief Title: Varenicline Treatment in Alcohol and Nicotine Dependent Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SUNY UMU IRBPHS #5656
Record Dates: First submitted 2008-07-28; First posted 2008-08-01 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Alcohol Dependence; Nicotine Dependence
Keywords: Varenicline; Smoking cessation; Schizophrenia; Schizoaffective disorder; Alcohol dependence; Nicotine dependence
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Alcoholism; Tobacco Use Disorder; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Varenicline (Active Comparator): Varenicline will be dispensed in 0.5 mg (blue capsules containing a 0.5 mg varenicline tablet) and 1 mg (red capsules containing a 1 mg varenicline tablet) capsules taken orally. During the first 3 days of medication, participants will take one blue capsule (0.5 mg tablet) of varenicline daily. If the medication is well-tolerated, the dose will be increased to one blue capsule (0.5 mg) po twice daily for 4 days. On day 8, the dose will be increased again to the standard dosing schedule of 1 red capsule (1 mg) po twice daily. At the end of the 8th week, varenicline will be discontinued.
  Interventions: Drug: Varenicline
- 2 Placebo (Placebo Comparator): Placebo will be dispensed in blue and red color coded capsules. During the first 3 days, participants will take one blue capsule po daily. If the medication is well-tolerated, the dose will be increased to one blue capsule po twice daily for 4 days. On day 8, the patients will take 1 red capsule po twice daily. At the end of the 8th week, placebo will be discontinued.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Varenicline will be dispensed in 0.5 mg and 1 mg tablets taken orally. During the first 3 days of medication, participants will take one 0.5 mg tablet of varenicline daily. If the medication is well-tolerated, the dose will be increased to 0.5 mg po twice daily for 4 days. On day 8, the dose will be increased again to the standard dosing schedule of 1 mg (1 tablet) po twice daily. At the end of the 8th week, varenicline will be discontinued.
  Other Names: Chantix
  Arms: 1 Varenicline
Drug: Placebo — Placebo will be dispensed in color-coded capsules. Blue capsules will contain 0.5 mg glucose (placebo), red capsules will contain 1 mg glucose (placebo).
  Arms: 2 Placebo

SUMMARY:
The aim of the proposed pilot study is to find out whether varenicline (ChantixTM) treatment decreases alcohol use and smoking in patients with schizophrenia or schizoaffective disorder. Varenicline may also improve cognition (memory and concentration) and negative symptoms (e.g. poor attention, poverty of speech, apathy, affective flattening, anhedonia) in patients with schizophrenia and comorbid nicotine and alcohol dependence.

DETAILED DESCRIPTION:
Alcohol use (more than 33%) and smoking (80-90%) commonly occur together in patients with schizophrenia. Varenicline (ChantixTM) has been approved by the FDA as a medication for smoking cessation. Recent animal studies have shown that chronic varenicline administration decreased alcohol consumption. There are no human data available on the effectiveness of varenicline in alcohol-use disorders.

The aim of the proposed pilot study is to find out whether varenicline treatment decreases alcohol use and smoking in patients with schizophrenia or schizoaffective disorder. Varenicline may also improve cognition (memory and concentration) and negative symptoms (e.g. poor attention, poverty of speech, apathy, affective flattening, anhedonia) in patients with schizophrenia and comorbid nicotine and alcohol dependence.

The proposed pilot study will enroll a cohort of up to 30 subjects with schizophrenia or schizoaffective disorder and nicotine and alcohol dependence, who are receiving ongoing outpatient mental health treatment from community providers. Subjects will be randomly assigned to one of the two treatment groups (varenicline vs. placebo). Following a one week screening phase, participants will be seen on day 4, day 8, then weekly over an 8-week treatment period. One week supply of medication will be dispensed at each study visit, with the exception of the first week, when only 4 days supply will be given on 2 days (visit 1 and 2). One month after discontinuation of medication, a follow-up interview will be conducted.

Varenicline and placebo will be dispensed in 0.5 mg and 1 mg color coded capsules. During the first 3 days of treatment, participants will take one 0.5 mg tablet of varenicline (or placebo) by mouth daily. If the medication is well-tolerated, the dose will be increased to 0.5 mg by mouth twice daily for 4 days. From day 8, the dose will be increased to the standard dosing schedule of 1 mg (1 tablet) by mouth twice daily. At the end of the 8th week, varenicline will be discontinued.

A structured clinical psychiatric interview and physical exam will be performed at baseline, along with a urine drug screen, which will be repeated on week 8, and at 1 month follow-up. Blood tests (complete blood count, basic metabolic panel, liver function tests) will be performed at baseline, then monthly.

During weekly study visits patients will undergo breath carbon-monoxide and breath alcohol testing, and they will answer questions about depression, smoking and alcohol use. Detailed assessment of psychiatric symptom severity (including neuropsychological testing) will be performed at baseline, at the end of the treatment phase (week 8). A functional MRI study will be performed at baseline and at the end of study to assess changes in blood flow, emotional processing and working memory related to varenicline treatment. In addition, genetic polymorphism of the α4β2 nicotinic acetylcholine receptor and gene expression changes related to drinking/smoking/psychosis and varenicline treatment will also be assessed.

The primary objectives of the proposed study are two fold: first to determine the feasibility of conducting a similar study on a larger scale, and second to establish pilot data for determining the effect size for hypothesized treatment effects on alcohol and nicotine use based on objective tests and self report. These estimates will help inform the minimum sample size needed for a larger future trial.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ages 18 to 69, with a DSM-IV diagnosis of Schizophrenia or Schizoaffective Disorder, receiving outpatient psychiatric treatment
* Currently taking antipsychotic medication for at least 4 weeks (medication is prescribed, compliance assessed based on self-report and collateral information)
* Current DSM-IV diagnosis of Nicotine Dependence
* Current DSM-IV diagnosis of Alcohol Dependence
* Subject expresses a desire to cut down or quit smoking and drinking (based on assessment with contemplation ladder)
* An average of at least one pack of cigarettes per day (>=20 cigarettes/day) over the 7 days prior to intake
* An average of at least 7 drinks over the 7 days prior to intake

Exclusion Criteria:

* Inability to give adequate informed consent
* Currently taking sustained - release bupropion (Zyban) or receiving any other form of bupropion, such as Wellbutrin or Wellbutrin SR; receiving another form of pharmacological smoking cessation treatment (e.g., nicotine gum or patch); or participating in another structured, formal smoking cessation program.
* Currently taking naltrexone (ReVia), Campral or Antabuse
* Participation in a clinical trial less than 3 months prior to intake
* History of suicide attempt in the past year
* History of hospitalization due to suicidal ideation in the past year
* Suicidal ideation at baseline
* Known allergic reaction to varenicline
* Female patients of childbearing potential who are sexually active, not sterile, and who deny using a form of birth control.
* Female patients who are pregnant or nursing.
* Significant unstable medical problems (e.g. impaired renal function).
* Significant unstable psychiatric disorders.
* Subjects who do not attend all required screening appointments.
* Subjects who have pending legal proceedings whose outcome may lead to incarceration within 3 months of intake.
* Positive urine drug screen for cocaine, opioids or amphetamine at baseline
* Current DSM-IV diagnosis of Cocaine, Opioid or Cannabis Dependence (1 month prior to enrollment)
* Metal implants or devices (e.g. aneurysm clips, cochlear implants, neural stimulators, cardiac pacemakers)
* Weight over 250 lbs
* Claustrophobia

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for alcohol use will be the number of drinks/week at the end of the treatment phase, relative to baseline and during-treatment data. | 8 weeks

SECONDARY OUTCOMES:
The outcome measure for smoking cessation effectiveness will be the amount of carbon monoxide in expired air at the end of the treatment phase, relative to data collected at baseline and during treatment. | 8 weeks
The safety of Varenicline use will be determined by examination of adverse events observed during the course of this investigation, with particular emphasis on comparing the frequency of adverse events in Placebo versus Treatment groups. | 8 weeks
Improvement in cognition will be assessed using the standardized California Verbal Learning Test (CVLT). | 8 weeks
Improvement in negative symptoms will be assessed using the PANSS negative score. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zsuzsa Szombathyne Meszaros, MD, PhD, Principal Investigator — SUNY Upstate Medical University, Department of Psychiatry; Steven L Batki, MD, Study Director — University of California, San Francisco
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Result] Meszaros ZS, Abdul-Malak Y, Dimmock JA, Wang D, Ajagbe TO, Batki SL. Varenicline treatment of concurrent alcohol and nicotine dependence in schizophrenia: a randomized, placebo-controlled pilot trial. J Clin Psychopharmacol. 2013 Apr;33(2):243-7. doi: 10.1097/JCP.0b013e3182870551. PMID 23422399
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273